CLINICAL TRIAL: NCT00799006
Title: A Phase 1 Placebo-Controlled Trial To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single Escalating Oral Doses Of PF-04620110 In Otherwise Healthy Overweight And Obese Subjects
Brief Title: A Single Dose Study Of PF-04620110 In Overweight And Obese, Otherwise Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B0961001
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Overweight
Keywords: Single Ascending Dose Study in Overweight subjects
MeSH Terms: conditions — Overweight | interventions — PF-04620110

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-04620110 (Experimental)
  Interventions: Drug: PF-04620110

INTERVENTIONS:
Drug: Placebo — Subjects will be given placebo or PF-04620110
  Arms: Placebo
Drug: PF-04620110 — A single oral dose of PF-04620110 will be given. The specific dose will depend on the cohort to which the subject is assigned and the period of the cross-over for that cohort. Initial planned doses are 0.3-30 mg but may be modified based on emerging PK and safety data.
  Arms: PF-04620110

SUMMARY:
PF-04620110 is a novel compound proposed for the treatment of Type 2 diabetes mellitus. The purpose of this study is to characterize the safety, tolerability, pharmacokinetics and pharmacodynamics following a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of approximately 27 to 35 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of PF-04620110 will be assessed by physical examinations, adverse event monitoring, 12 lead ECGs, continuous cardiac monitoring over the first 8 hours after dosing, vital sign and clinical safety laboratory measurements. | 4 days/dose group
The single dose pharmacokinetics of PF-04620110 will be assessed | 4 days/dose group

SECONDARY OUTCOMES:
Secondary pharmacodynamic endpoints will include postprandial lipid metabolism measures | 1 day/dose group

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Amin NB, Saxena AR, Somayaji V, Dullea R. Inhibition of Diacylglycerol Acyltransferase 2 Versus Diacylglycerol Acyltransferase 1: Potential Therapeutic Implications of Pharmacology. Clin Ther. 2023 Jan;45(1):55-70. doi: 10.1016/j.clinthera.2022.12.008. Epub 2023 Jan 21. PMID 36690550
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961001&StudyName=A%20Single%20Dose%20Study%20Of%20PF-04620110%20In%20Overweight%20And%20Obese%2C%20Otherwise%20Healthy%20Volunteers